CLINICAL TRIAL: NCT04276727
Title: A Phase II RCT of Topical Menthol Gel Versus Placebo in the Treatment of Chemotherapy Induced Peripheral Neuropathic Pain
Brief Title: Menthol In Neuropathy Trial
Acronym: MINT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MINT
Record Dates: First submitted 2019-11-08; First posted 2020-02-19 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy
Keywords: CIPN; Peripheral neuropathy; Chemotherapy; Neuropathic pain
MeSH Terms: conditions — Peripheral Nervous System Diseases; Neuralgia

STUDY DESIGN:
Intervention Model Description: Randomised, double-blind placebo controlled
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Gel tubes will be supplied with similar labelling, identified by blinded drug pack numbers which can be linked to the treatment allocation if an emergency need arises. The menthol and placebo gels have a similar blue colour and both have a minty odour.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Menthol (Active Comparator): Menthol gel to be applied twice a day for 6 weeks - toes to knees, fingertips to elbows, top and base of spine.
  Interventions: Drug: MINT study IMP
- Placebo (Placebo Comparator): Placebo gel to be applied twice a day for 6 weeks - toes to knees, fingertips to elbows, top and base of spine.
  Interventions: Drug: MINT study IMP

INTERVENTIONS:
Drug: MINT study IMP — Application of gel for 6 weeks.

SUMMARY:
Patients will be recruited who have peripheral neuropathy due to chemotherapy. They will be given a blinded treatment of gel containing either menthol (3%) or placebo to be applied for 6 weeks, twice a day. Assessments of pain, neuropathic symptoms and impact on quality of life will be done at baseline, 6 weeks and 12 weeks. Functional magnetic resonance imaging (fMRI) scans will be done at baseline and 6 weeks. Physical activity data will also be collected to be analysed in conjunction with pain assessments.

DETAILED DESCRIPTION:
Modern cancer treatments, while more effective at prolonging life, are associated with some long lasting effects, especially nerve pain. This occurs in up to 90% of patients and 50% of patients still experience nerve pain a year after treatment. Not only is this distressing in itself but the investigators now understand that this treatment-related pain is exacerbating other pains, making cancer pain more difficult to control. The problem with managing nerve pain caused by treatment is that there is no predictable and effective treatment.

Our team has discovered that menthol cream or gel applied to the skin in the area of nerve pain can be effective. This trial seeks to provide better evidence of using this simple, cheap, non-toxic treatment. Participants will be given either menthol gel to the affected area or a placebo gel which smells, looks like and has the same texture as menthol but has no active drug. The gel will be applied twice a day for 6 weeks.

Participants will initially be assessed for pain and its impact on function, mood and quality of life and, if possible, will also have an fMRI scan immediately before starting menthol treatment and after 6 weeks of treatment. They will also have some assessments a further 6 weeks after treatment finishes. As part of impact on function assessment, participants will be asked to wear a physical activity monitor for a few days prior to each of the three main assessment points.

Our group has used special scans of the brain called fMRI to help identify if a treatment has real potential for patients. Sometimes, in early studies of a new treatment, patients can believe that the treatment has a real effect, but in fact it is a placebo effect. FMRI scans in this study will help to identify if menthol gel is having a true pain relieving effect, by comparing the patient's reports of pain with their scan findings. This will be very helpful in aiding the decision of how the research team conduct any future larger clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Patients have received any neurotoxic chemotherapy.
2. Patients have experienced post treatment Chemotherapy Induced Peripheral Neuropathy (CIPN) pain for a minimum of 3 months after completing chemotherapy.
3. Patients reporting a distressing or uncomfortable neuropathic symptom (such as pain or tingling) with an average score in the last 24 hours of ≥5 on a scale of 0-10 with 0 being none, according to the Numeric Rating Scale for pain.
4. Aged 18 years or over at study entry.
5. Patient's Oncology team agrees to their taking part in the study.
6. Patients are able to provide written informed consent to participation in the study after explanation of the study protocol.
7. In the opinion of the investigator, the patient is able to complete the various assessments.
8. Neuropathy must be confined to the distal extremities (distal to elbows and/or knees).

Exclusion Criteria:

1. Pre-existing or history of peripheral neuropathy due to any cause other than chemotherapy (diabetes, alcohol, toxin, hereditary, etc.).
2. Patients with any contraindication to the use of topical therapy or menthol.
3. Neurological conditions which may influence findings (such as Multiple Sclerosis or residual signs/symptoms from a previous stroke).
4. Skin conditions which prevent assessment of the relevant areas affected by peripheral neuropathy.
5. Suffering from significant psychiatric illness, which would hinder their completion of the study in the opinion of the investigator.
6. General medical condition is unstable or rapidly deteriorating, such that they are unlikely to be able to contribute to the study.
7. In the opinion of the Research Team or their usual medical team, would be unable to complete the study protocol for any other reason.
8. Current treatment of ≤ 30 days duration with topical lidocaine patch/gel or anticonvulsants, tricyclic antidepressants, MAO inhibitor, or other neuropathic pain medication agents such as carbamazepine, phenytoin, valproic acid, gabapentin/pregabalin, lamotrigine or amifostine. (If on the same dose of any of these medications for >31 days, patients will be asked to continue these for the duration of the study. Analgesic agents such as acetaminophen, nonsteroidal anti-inflammatory agents, or opioids, are allowed if on the same doses for >31 days).
9. Application of capsaicin cream or patch (to the limb extremities) currently or within the last 30 days (as this would interfere with application of the menthol gel and potentially study outcome).
10. Patients with significant pain other than CIPN (ie pain worse than the CIPN).
11. Other medical conditions, which in the opinion of the treating physician/allied health professional would make this protocol unreasonably hazardous for the patient.
12. Participants previously randomised into this study.
13. Participants not prepared to stop using any other physical activity meter.
14. Co-enrolment in any other pain treatment studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2022-03-24 (Actual); Study Completion 2022-03-24 (Actual)

PRIMARY OUTCOMES:
Reduction in CIPN symptoms | 6 weeks
  A clinically significant reduction in pain (at least a 30% decrease in total BPI SF score as relates to the index neuropathic pain) between baseline and 6 weeks.

SECONDARY OUTCOMES:
Treatment effect on Chemotherapy Induced Peripheral Neuropathy | 6 weeks
  Changes in EORTC QLQ (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaires) CIPN-20 (severity of 20 symptoms rated on 4 point scale from Not at all to Very much)
Treatment effect on quality of life functions | 6 weeks
  Changes in EORTC QLC-c30 scores (30 symptoms on same scale as CIPN)
Treatment effect on pain scores | 6 weeks
  Changes in Brief Pain Inventory - Short Form scores (13 symptoms rated from 0 None to 10 Worst)
Treatment effect on anxiety and depression | 6 weeks (14 symptoms rated from 0 to 3 in severity)
  Changes in Hospital Anxiety and Depression Scale (HADS) scores
Treatment effect on pain catastrophisation | 6 weeks (13 questions rated from 0-4 in severity)
  Changes in Pain Catastrophising Scale (PCS) scores
Treatment effect on side effects | 6 weeks
  Changes in side effects (Yes/No to any SEs, description of SE to be given)
Treatment effect on physical activity | 6 weeks
  Changes in Actigraph data (measures of step counts, amount of moderate/vigorous activity and sleep times/efficiency)
Perceived effects of IMP | 6 weeks
  Changes in perceived effects questions (How long participant thinks treatment takes to take effect and how long it lasts for)

OTHER OUTCOMES:
Changes in Functional Magnetic Imaging data | 6 weeks
  Changes in FMRI data pre and post treatment
Post treatment changes in CIPN | 12 weeks (from baseline)
  Changes in CIPN-20 scores (see secondary outcomes above for details of all questionnaire measures)
Post treatment changes in quality of life measures | 12 weeks (from baseline)
  Changes in QLQ-c30
Post treatment changes in pain scores | 12 weeks (from baseline)
  Changes in BPI-SF
Post treatment changes in anxiety and depression | 12 weeks (from baseline)
  Changes in HADS scores
Post treatment changes in pain catastrophising | 12 weeks (from baseline)
  Changes in PCS
Post treatment changes in side effects | 12 weeks (from baseline)
  Changes in Side effects
Post treatment changes in physical activity | 12 weeks (from baseline)
  Changes in Actigraph data
Changes in sensory measures | 6 weeks and 12 weeks (from baseline)
  Changes in QST data

CONTACTS AND LOCATIONS:
Locations (1):
- Western General Hospital, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Anyone interested in secondary analysis of the data should contact the Chief Investigator in the first instance.